CLINICAL TRIAL: NCT05715554
Title: Community-based Individualized Homeopathic Rehabilitation in Post COVID-19 Patients: Results of a Pilot, Pragmatic, Randomized, Open Label, Controlled Trial Investigating Acceptability and Feasibility
Brief Title: Community-based Individualized Homeopathic Rehabilitation in Post COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innowage Limited (Industry)
Collaborators: Gyansanjeevani India (Unknown); Collaborative Homeopathy Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-G-001
Record Dates: First submitted 2023-02-06; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Post-COVID Syndrome
Keywords: Rehabilitation; Homeopathy; Post-COVID Syndrome
MeSH Terms: interventions — Homeopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homeopathy Group (Experimental): Individualized Homeopathy Treatment provided by homeopathic physicians
  Interventions: Other: Homeopathy
- Standard Group (No Intervention): Usual care provided by primary care physicians were followed by patients in the standard group

INTERVENTIONS:
Other: Homeopathy — Individualized homoeopathic medicines on impregnated lactose pellets was prescribed based on totality of physical, emotional, and mental symptoms.
  Arms: Homeopathy Group

SUMMARY:
A growing number of studies identify a spectrum of persistent symptoms experienced by COVID-19 patients for months after recovery. Symptoms include cough, fatigue, dyspnea, pain, and brain fog (cognitive impairment, including confusion and memory loss), which have a negative impact on daily activities. Homoeopathic practitioners from around the world have documented a number of successful cases of Post COVID treatment. Even though evidence from practice-based research is limited, the purpose of the current study was to evaluate the effect of individualized homoeopathy treatment on post-COVID syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 history
* Persistent respiratory symptoms for more than three months after COVID-19
* Able to provide informed consent

Exclusion Criteria:

* Presence of respiratory issues without COVID-19 diagnosis
* On complementary and Alternative Treatment
* Symptoms of infection
* Pregnancy or Breastfeeding
* Cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Cough severity | 8 weeks
  Severity from 0-10 visual analog scale, where 0 is none to 10 is most severe.

SECONDARY OUTCOMES:
Change in dyspnea | 8 weeks
  Change in dyspnea using Modified Borg Scale (0 is best to 10 is wore)
Change in Fatigue | 8 weeks
  Change in fatigue severity scale (0 -7 no fatigue to worse )
change in Quality of Life | 8 weeks
  Saint George Respiratory Questionnaire (SGRQ)to assess the quality of life (scores ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Sadhana Sharma, Principal Investigator — Gyansanjeevani India; Vesna Marinković, Study Director — Collaborative Homeopathy Research Network; Neha Sharma, Study Chair — Innowage Limited
Locations (5):
- India (5):
  - Gyansanjeevani India, Dausa, Rajasthan
  - Gyansanjeevani India, Jaipur, Rajasthan
  - Gyansanjeevani India, Mandāwa, Rajasthan
  - Gyansanjeevani India, Sawai Madhopur, Rajasthan
  - Gyansanjeevani India, Sīkar, Rajasthan